CLINICAL TRIAL: NCT07219537
Title: Pilot Study for Imaging the Lower Gastrointestinal Tract Using a Retro-TCE Capsule
Brief Title: A Study for Imaging the Lower Gastrointestinal Tract Using a Retro-TCE Capsule
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2022P001154
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Lynch Syndrome; Crohn Disease; Inflammatory Bowel Diseases; Healthy
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Healthy (Experimental): 20 healthy adult participants with no pre-existing gastrointestinal disorders will be enrolled at MGH.
  Interventions: Device: Feasibility of using an OCT-based Retrograde Tethered Capsule Endomicroscope device to image the lower GI tract
- With Disease (Experimental): 10 adult participants with a confirmed diagnosis of Lynch Syndrome, Crohn's Disease, or Inflammatory Bowel Disease will be enrolled at MGH.
  Interventions: Device: Feasibility of using an OCT-based Retrograde Tethered Capsule Endomicroscope device to image the lower GI tract

INTERVENTIONS:
Device: Feasibility of using an OCT-based Retrograde Tethered Capsule Endomicroscope device to image the lower GI tract — 30 participants will be enrolled in this study. All consented participants will receive the same intervention.

SUMMARY:
The investigators have developed an inexpensive tool to take pictures in the lower GI tract without sedation and to look for signs of disease. The tool is a capsule, about the size of a fish oil or multi-vitamin supplement, attached to a string. The capsule and string are connected to a motor to allow the capsule to advance up the participant's lower GI tract. The capsule will be inserted into the participant's lower GI tract and advance upward via a slow spiral motion. The capsule is connected to an imaging system that saves and displays the images in real time.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older.
* Are healthy or with a confirmed diagnosis of Lynch Syndrome
* Are capable of giving informed consent.
* Are able to follow bowel prep instructions
* Had a colonoscopy 0-24 months prior that did not show any abnormalities or individuals who report no gastrointestinal symptoms and no knowledge of any lower GI tract disease or abnormality and volunteer through Rally.

Exclusion Criteria:

* Who are over 75 years of age or older
* With a history or current diagnosis of colonic and/or anal strictures
* With a current diagnosis of any bleeding disorders
* Who currently use drugs that interfere with coagulation (excluding low-dose aspirin)
* With a history or current diagnosis of colorectal cancer
* With a history or current diagnosis of diverticulosis or diverticulitis
* With any prior anorectal, colorectal, or colonic surgery
* With a history of volvulus or torsion
* Who are pregnant
* With contraindications to bowel prep or colonoscopy
* With severe acute inflammatory bowel disease
* With large hemorrhoids or hemorrhoidal bleeding or banding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ability of the R-TCE capsule to acquire quality images of the lower GI tract | Imaging data is collected during the study procedure and analyzed within one year of collection.

SECONDARY OUTCOMES:
Tolerability of the R-TCE Capsule in an unsedated participant | Day 1
  R-TCE imaging will be conducted in unsedated participants. The study team will ask the participants about their comfort level throughout the procedure. Participants will be asked to score the tolerability of the procedure using a scoring system from 0 to 10. With 0 being the most tolerable to10 being the least.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States